CLINICAL TRIAL: NCT02442739
Title: A Randomized, Double Blind, Feasibility Study of Oral Ketamine Versus Placebo for Prevention of Depression in Patients Undergoing Treatment for Pancreatic or Head and Neck Cancers
Brief Title: Ketamine for Preventing Depression in Patients Undergoing Treatment for Pancreatic or Head and Neck Cancers
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI voluntary closure due to low accrual
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Scott A. Irwin, MD, PhD, Associate Professor, Psychiatry & Behavioral Neurosciences, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IIT2015-22-IRWIN-KETPREVE; 1R21CA197023-01A1 (NIH)
Record Dates: First submitted 2015-05-07; First posted 2015-05-13 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Cancer; Pancreatic Cancer; Depression
Keywords: Ketamine; Prevention of depression
MeSH Terms: conditions — Head and Neck Neoplasms; Pancreatic Neoplasms; Depression | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): oral ketamine 0.5 mg/kg mixed with syrup
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): oral placebo (syrup)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine 0.5 mg/kg mixed with syrup will be given by mouth once a week for 12 weeks.
  Other Names: Ketalar
  Arms: Ketamine
Other: Placebo — Placebo syrup will be given by mouth once a week for 12 weeks.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to see if it is safe to give patients with pancreatic or head and neck cancer a low dose of the FDA approved anesthetic drug ketamine at the same time they receive radiation and/or chemotherapy for their cancer treatment to prevent depression and its effects. Researchers would also like to see if giving ketamine at the same time as cancer treatment is practical and reasonably acceptable to the patient.

New onset depression is highly frequent in those with head and neck cancer, and depression has many negative consequences for outcomes in those patients. Depression has been known to have greater incidence in pancreatic cancer patients than in patients with other malignancies.

Therefore, investigators would also like to see if giving patients ketamine during their routine cancer treatment will prevent the onset of depression and its negative effects on cancer treatment outcomes, and also help with anxiety, pain, and quality of life. The study will also use a placebo to compare to the good and/or bad effects of ketamine. A placebo is not an active drug and it will be look the same as ketamine, as a liquid to be taken by mouth.

Ketamine is approved by the U.S. Food and Drug Administration (FDA) as a general anesthetic by itself for some diagnostic and surgical procedures or combined with other general anesthetic agents. It has also been shown to reduce cancer pain. Ketamine is considered experimental in this study because it is not approved by the FDA for the prevention of depression.

DETAILED DESCRIPTION:
This is a prospective, single center, double blind, randomized, two-arm feasibility study of oral ketamine versus placebo for the prevention of depression in non-depressed patients with head and neck or pancreatic cancer undergoing curative intent cancer therapy. Approximately 40 patients with head and neck cancer or pancreatic cancer about to undergo cancer therapy will be randomized 1:1 to receive study treatment with one of the following regimens:

* Arm A: weekly oral administration of 0.5 mg/kg ketamine
* Arm B: weekly oral administration of placebo

Consenting patients will undergo screening procedures, and if eligible, a baseline interview and brief questionnaires regarding depression, mental and emotional health, and quality of life assessments.

Study treatment will be administered for 12 weeks unless the patient experiences unacceptable toxicities, exhibits moderate to severe depressive symptoms, or withdraws consent. Patients on the placebo treatment arm will not be eligible to cross over to the ketamine arm at evidence of depression but will be removed from the study and treated with standard medical management for depression.

Patients will be asked to complete psychosocial measurements every two weeks, before study medication/placebo administration, while on study treatment and monthly during a five-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent.
2. Stage -II-IV epidermoid cancer of the head and neck OR stage III-IV pancreatic cancer, with prognosis of at least three months, per oncologist.
3. Within two weeks of starting or from having started, curative intent therapy for head and neck cancer.
4. Age ≥ 18 years.
5. Adequate liver function as defined by:

   * ALT < 5 X institutional upper limit of normal (ULN)
   * AST < 5 X institutional ULN
   * Total bilirubin < 5 X institutional ULN
6. Both men and women of all races and ethnic groups are eligible for this trial.
7. Use of antidepressants is permitted if dose has been the same for at least 12 weeks prior to study entry if patient still DOES NOT meet exclusion criteria #3.
8. Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform the study team and her treating physician immediately. Urine pregnancy testing will be done throughout the trial for women of childbearing potential.
9. Must read and understand English fluently.

Exclusion Criteria:

1. Receiving another investigational agent on a clinical trial that prohibits participation in other studies of investigational agents.
2. Meets Mini International Neuropsychiatric interview (MINI) criteria for major depression, schizophrenia, bipolar illness, delirium or psychosis.
3. Has moderate to severe depression according to both the Quick Inventory of Depressive Symptomatology-Self Rated 16 (QIDS-SR-16) score of ≥ 11 AND a Hospital Anxiety and Depression Scale (HADS) Depression subscale score of ≥ 8.
4. Has Suicidal Risk Assessment (SRA) scores ≥ 6.
5. Use of monoamine oxidase inhibitors within 14 days of study entry.
6. Diagnosed with melanoma or lymphoma cancer of the head and neck.
7. Diagnosed with Stage I or II pancreatic cancer or with anticipated survival of less than three months.
8. History of allergic reactions or hypersensitivity to ketamine.
9. Severe cardiac insufficiency (NYHA III or IV), with uncontrolled and/or unstable cardiac or coronary artery disease.
10. History of significant tachyarrhythmia, severe angina, or myocardial ischemia
11. Poorly controlled hypertension (Systolic Blood Pressure > 180 mmHG or Diastolic Blood Pressure > 100 mmHG), with or without antihypertensives.
12. If a woman is or becomes pregnant or is nursing at any time before or during the treatment period, she will be excluded from the study.
13. Score of ≥ 8 on the WHO Alcohol Use Disorders Identification Test (AUDIT, sensitivity of 0.8).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients pre-screened that were potentially eligible for study participation. | 36 months
Proportion of patients that were potentially eligible who were approached. | 36 months
Proportion of approached patients that decline study participation and why. | 36 months
Proportion of approached patients that agreed to participate. | 36 months
Proportion of approached that were randomized. | 36 months
Proportion of patients discontinuing prematurely from study treatment for any reason, including side effects attributed to ketamine or side effects attributed to placebo, documenting reasons for dropout. | 36 months
Proportion of patients that are evaluable | 36 months
  Subjects with a baseline and one post-baseline visit are evaluable and will be included in the analyses.

SECONDARY OUTCOMES:
Treatment-related adverse events | 4 months
  Adverse Events rated as possibly/probably related to study treatment
Patient-reported tolerability questionnaire (FIBSER) | 4 months
Treatment expectancy and satisfaction as measured by the credibility/expectancy questionnaire (CEQ). | 4 months

OTHER OUTCOMES:
Incidence of new onset mild, moderate, or severe depressive symptoms as assessed by questionnaire (QIDS-SR-16) | 4 months
Depression-free survival | 4 months
Severity of cancer-related pain as assessed by a visual analog scale (VAS) | 4 months
Anxiety and depressive symptoms as assessed by questionnaire (HADS) | 4 months
Quality of life as assessed by questionnaire (UW-QOL) | 4 months
Suicide risk and ideation as assessed by questionnaire (SRA) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott Irwin, MD, PhD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States